CLINICAL TRIAL: NCT01926873
Title: MULTI-CENTER COGNITION ASSESSMENT IN HEALTHY SUBJECTS TO COLLECT REFERENCE DATA FOR COMPARISON TO PATIENTS WITH DEPRESSION
Brief Title: A Screening Study To Assess The Cognition Status in Healthy Volunteers
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: BP28865; 2013-001261-16 (EudraCT Number)
Record Dates: First submitted 2013-08-16; First posted 2013-08-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Samples

GROUPS / COHORTS (1):
- Healthy volunteers

SUMMARY:
This multi-center screening study will conduct a cognition assessment to collect reference data for comparison to patients with depression in healthy volunteers. Data will be collected for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, 18 to 65 years of age, inclusive
* Healthy volunteers with a stable chronic disease that is not associated with cognitive deficits (e.g. asthma) and does not require any treatment known to affect cognition have to be discussed with the medical monitor before enrollment
* A body mass index between 18 to 30 kg/m2 inclusive
* Able to participate and willing to give written informed consent and to comply with the study restrictions
* At least second generation resident in the country of origin

Exclusion Criteria:

* Current or past history of a psychiatric disorder
* Family history of psychiatric disorders
* Suspicion or evidence of regular consumption of drugs of abuse or a positive drug test at the screening visit
* Acute or chronic disorder which is not stable or may affect cognition or needs treatment affecting cognition
* Change of smoking behavior or smoking cessation therapy within 30 days before screening visit
* Positive result on hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) 1 and 2
* Systolic blood pressure greater than 140 or less than 90 mm Hg, and diastolic blood pressure greater than 100 or less than 50 mm Hg
* Resting Pulse Rate greater than 100 or less than 45 beats per minute
* Clinically significant abnormalities in laboratory test results or in ECG assessment at screening visit
* Participation in an investigational drug study within 1 month prior to baseline

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2013-08; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Cognitive status of volunteers | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (12):
- United States (5):
  - San Diego, California
  - Atlanta, Georgia
  - Oak Brook, Illinois
  - Cedarhurst, New York
  - Salt Lake City, Utah
- Germany (4):
  - Freiburg im Breisgau
  - Mainz
  - Mannheim
  - Schwerin, Mecklenburg-Vorpommern
- Poland (3):
  - Bialystok
  - Choroszcz
  - Tuszyn